CLINICAL TRIAL: NCT07052864
Title: Efficacy of Dexamethasone in Preventing Postspinal Hypotension in Elderly Patients Undergoing Orthopedic Surgery: a Randomized Controlled Study
Brief Title: IV Dexamethasone in Preventing Post Spinal Hypotension
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Muhammad Haroon Anwar, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: F.5-2/2024(ERRC)/PIMS
Record Dates: First submitted 2025-06-29; First posted 2025-07-07 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Hypotension During Surgery
MeSH Terms: interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Intervention Model Description: After taking informed consent participants will be divided into two equal groups using computer generated random numbers. The participants in group D will receive 8 mg of IV Dexamethasone in 100ml Normal saline 1 hour before induction of spinal anesthesia while participants in group C will receive 100ml of Normal saline 1 hour before induction of spinal anesthesia. 1 hour after administration of IV Dexamethasone or placebo patient will be brought into OR, ASA monitoring will be attached, Sub Arachnoid block will be induced with 15mg of hyperbaric bupivacaine, patient will be made to lie down, level of block will be assessed and surgery will be started. Intraoperatively hemodynamics will be recorded at 5 minutes interval for first 30 minutes. Any fall in blood pressure by more than 20% from baseline will be noted and treated with Phenylephrine IV bolus.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group Dexamethasone (Experimental): Participants entering this arm of Parallel randomized control trial will receive 8mg of IV Dexamethasone in 100ml Normal saline 1 hour before induction of spinal anesthesia.
  Interventions: Drug: Dexamethasone
- Group Placebo (Placebo Comparator): Participants entering this arm of Parallel randomized control trial will receive 100ml Normal saline 1 hour before induction of spinal anesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 8 mg of Intravenous Dexamethasone in 100 ml Normal saline given 1 hour before anesthesia induction
  Arms: Group Dexamethasone
Drug: Placebo — 100ml of Normal saline administration 1 hour before anesthesia induction
  Other Names: Normal Saline
  Arms: Group Placebo

SUMMARY:
Orthopedic lower limb procedures are carried out under spinal anesthesia which involves administration of drugs in the space surrounding the spinal cord. From there the drug acts on the spinal cord blocking electrical signals moving across nerve fibers thereby providing sufficient pain relief and surgical conditions. However blocking of these fibers result in reduce signal transmission to blood vessels and heart resulting in fall in blood pressure. Various drugs can be used to treat or prevent this hypotension. One such drug is Dexamethasone which is a steroid. This drug can be administered before spinal anesthesia through Intravenous route to prevent fall in blood pressure.

DETAILED DESCRIPTION:
Lower limb orthopedic surgeries are carried out under Sub Arachnoid block which is associated with sympathectomy resulting in vasodilation and hypotension. The hypotension can compromise end organ perfusion and pre-disposes the person to end organ damage such as Myocardial infarction, stroke and renal injury. Therefore treatment and prevention of post spinal hypotension is one of the major goals to improve peri-operative outcomes. One such drug which can be used to prevent post spinal hypotension is Dexamethasone which can be given prophylactically to prevent post spinal hypotension as the drug causes increase in systemic vascular resistance thereby counteracting post spinal vasodilation and hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthopedic surgery under spinal anaesthesia.
* ASA I & II.

Exclusion Criteria:

* Known case of ischemic heart disease.
* Patients having contraindication to spinal anesthesia (e.g.- coagulopathy, thrombocytopenia, allergy to local anesthetic agent).
* Patients using corticosteroids or drugs that affect serotonin (e.g., selective serotonin reuptake inhibitor).
* Patients with uncorrected hypovolemia.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | baseline, 5 mins, 10 mins, 15 mins, 20 mins, 25 mins,30 mins
  This is the highest blood pressure during cardiac cycle occurring at the peak of systole measured by Non invasive automated blood pressure cuff
Diastolic Blood Pressure | baseline, 5 mins, 10 mins, 15 mins, 20 mins, 25 mins,30 mins
  This is the lowest blood pressure during cardiac cycle measured by Non invasive automated blood pressure cuff
Mean Blood Pressure | baseline, 5 mins, 10 mins, 15 mins, 20 mins, 25 mins,30 mins
  This is the average blood pressure during cardiac cycle measured by Non invasive automated blood pressure cuff

SECONDARY OUTCOMES:
Number of Hypotensive episodes | Intraoperative period
  This will be the number of times in the intraoperative period the patient experience fall in either systolic, diastolic or mean blood pressure by more than 20% from baseline
Rescue Phenylephrine | Intraoperative period
  This will be the total amount of phenylephrine administered in intraoperative period to the patient in case of fall in either systolic, diastolic or mean blood pressure by more than 20% from baseline
Rescue intravenous fluid | Intraoperative period
  This will be the total amount of IV crystalloid fluid administered in intraoperative period to the patient in case of fall in either systolic, diastolic or mean blood pressure by more than 20% from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Anesthesia and Critical Care Medicine, Pakistan Institute of Medical Sciences, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashoor TM, Hussien NS, Anis SG, Esmat IM. Dexamethasone blunts postspinal hypotension in geriatric patients undergoing orthopedic surgery: a double blind, placebo-controlled study. BMC Anesthesiol. 2021 Jan 11;21(1):11. doi: 10.1186/s12871-021-01232-w. PMID 33430772
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33430772/